CLINICAL TRIAL: NCT05744193
Title: Comparison of Multinutrient Human Milk Fortifiers in Preterm Infants: A Non-inferiority Single-blind, Randomized Controlled Trial (RCT)
Brief Title: Feeding Study in VLBW Premature Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3394-1
Record Dates: First submitted 2023-01-31; First posted 2023-02-24 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: VLBW - Very Low Birth Weight Infant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Commercial Liquid Human Milk Fortifier (Active Comparator): Liquid human milk fortifier to be added to human milk
  Interventions: Other: Exempt Infant Formula
- Liquid Human Milk Fortifier - Standard Protein (Experimental): Liquid human milk fortifier to be added to human milk
  Interventions: Other: Exempt Infant Formula
- Liquid Human Milk Fortifier - High Protein (Experimental): Liquid human milk fortifier to be added to human milk
  Interventions: Other: Exempt Infant Formula

INTERVENTIONS:
Other: Exempt Infant Formula — Liquid human milk fortifier to be added to human milk daily

SUMMARY:
A multi-center, single-blind, randomized, controlled, parallel-designed, prospective trial to compare growth between preterm infants fed one of three study human milk fortifiers added to human milk

ELIGIBILITY:
Inclusion Criteria:

* Clinically and metabolically stable
* Birth weight 700 g to less than or equal to 1,250 g
* Appropriate birth weight for gestational age
* 24 0/7 to 32 0/7 weeks' gestational age at birth
* Exclusively fed human milk
* Signed informed consent and authorization to use and/or disclose PHI

Exclusion Criteria:

* Metabolic or chronic disease
* 5-minute Apgar score <4
* Major surgery
* Ventilator dependent
* Fluid restriction
* Grade III or IV intraventricular hemorrhage (IVH)

Ages: 168 Days to 224 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Weight gain | Daily for 28 days
  grams/kg/day

SECONDARY OUTCOMES:
Feeding Tolerance | Daily for 28 days
  Achievement of full enteral feeding, incidence of (TPN, Bloody stools, Feeding interruptions, Drop in feeding volume)
Rate of Length and head circumference gain | weekly up to day 28
  cm/week
Total energy intake | 28 days
  kcal
Total protein intake | 28 days
  grams
Respiratory status | 28 days
  Incidence of Apnea, Bradycardia, Supplemental oxygen/Continuous positive airway pressure/Nasal cannulation, Mechanical ventilation
Incidence of NEC | Study Day 0 through 28
  Modified Bell's Staging Criteria
Incidence of sepsis - clinical symptoms | Study Day 0 through 28
  Clinical symptoms - Changes in respiration, blood pressure, body temperature, stool, blood sugar and heart rate
Incidence of sepsis - culture for pathogens | Study day 0 through 28
  Culture for pathogens - no culture, culture-negative, culture-positive, presumed contaminant
Incidence of sepsis - Antibiotic use | Study Day 0 through 28
  Antibiotic use duration - less than 5 days ; 5 days or more
Total serum CO2 | Study days 0, 14, 28
  less than 18 mmol/L
Metabolic Acidosis | Study days 0, 14, 28
  If CO2 <18 mmol/L then Blood gas; Acidity (pH), Carbon dioxide, partial pressure (pCO2; torr), Bicarbonate (mmol/L); Base Excess (mmol/L)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Augusta University, Augusta, Georgia
  - Riley Children's Hospital, Indianapolis, Indiana
  - NYU Langone Hospital, Long Island, Mineola, New York
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Weill Cornell Medicine, New York, New York